CLINICAL TRIAL: NCT04294446
Title: Post-market Study of the Biodesign® Hernia Graft
Brief Title: Post-market Study of the Biodesign Hernia Graft
Status: Recruiting | Type: Observational
Sponsor: Cook Biotech Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-004
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Biodesign Hernia Graft — The Biodesign Hernia Graft is comprised of 8 layers of decellularized porcine small intestinal submucosa (SIS) that has been pressed-lyophilized (i.e., freeze-dried under vacuum pressure) to laminate the component sheets (i.e., layers) together. In addition, it is perforated and sewn with 4-0 Trisorb suture (polyglycolic acid (PGA); Samyang Corporation, Seoul, South Korea). The suture is distributed in a diamond pattern across the graft and along the periphery and is intended to mitigate delamination of the layers upon rehydration and/or manipulation during implantation. Being a completely biologic device, the Biodesign Hernia Graft is considered MR safe.

SUMMARY:
The purpose of this study is to collect data on the performance of the Biodesign® Hernia Graft when used to reinforce soft tissues during ventral hernia repair.

DETAILED DESCRIPTION:
This multicenter, open-label, prospective clinical study will evaluate the performance of the Biodesign Hernia Graft to reinforce soft tissues during ventral hernia repair.

This post-market study will enroll up to 95 patients at up to 10 clinical sites. Each clinical site will be limited to a maximum of 50 patients to ensure a variety of patients and surgical techniques are represented. There is no minimum enrollment number per site.

This study has been designed as a multicenter, open-label, prospective study to collect data on the performance of the Biodesign Hernia Graft. The inclusion and exclusion criteria for this study have been selected based on the instructions outlined in the IFU so that the results from this study can provide data on the real-world use of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Primary or recurrent ventral hernia in need of surgical repair utilizing a Biodesign Hernia Graft

Exclusion Criteria:

1. Known sensitivity to porcine material

   For the study, the following patients will also be excluded:
2. Age < 18 years
3. Unable or unwilling to provide informed consent
4. Life expectancy of less than one year from the date of the index procedure
5. Patients will be excluded from the study if they never receive a Biodesign Hernia Graft during their index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet all of the inclusion criteria and none of the exclusion criteria will be invited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | 1-year
  Hernia recurrence through 1-year follow-up

SECONDARY OUTCOMES:
Device-, procedure-, and hernia-related adverse event rates | 2-year
  Summarize the adverse event rates for normal commercial use of the device (e.g., seroma and infection rates)
Hernia recurrence rate through 2-year follow-up | 2-year
  Assess the long-term success of the device in the reinforcement of hernia repairs through 2-year follow-up
Operative times | 2-year
  What was the operation time for the ventral hernia repair?
Hospital stay | 2-year
  Duration of hospital stay
Hospitalization times for related Serious Adverse Events (SAEs) | 2-year
  What was the hospitalization times for any related SAEs?
Patient-reported quality of life: questionaire | 2-year
  Patient-reported quality of life assessed by completion of a questionaire

CONTACTS AND LOCATIONS:
Locations (3):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No